CLINICAL TRIAL: NCT00955682
Title: Persistence of Antibodies After GSK Biologicals' Meningococcal Vaccine GSK134612 in Toddlers
Brief Title: Study to Evaluate Persistence of Antibodies After Vaccination With Meningococcal Vaccine GSK134612
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112036; 2008-003824-51 (EudraCT Number)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal vaccine GSK134612
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Group A (Experimental): Subjects who received GSK vaccine 134612 in the primary vaccination study 109069 and will be boosted 4 years after primary vaccination with the same meningococcal vaccine as given in the primary study.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Group B (Active Comparator): Subjects who received Meningitec™ vaccine in the primary vaccination study 109069 and will be boosted 4 years after primary vaccination with the same meningococcal vaccine as given in the primary study.
  Interventions: Biological: Meningitec™

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One intramuscular dose (Booster)
  Arms: Group A
Biological: Meningitec™ — One intramuscular dose (Booster)
  Arms: Group B

SUMMARY:
Subjects were previously vaccinated at 12 to 23 months of age. This extension study starts 24 months after vaccination and the subjects who were vaccinated in the primary study will be enrolled in this extension phase. No new subjects will be enrolled.

DETAILED DESCRIPTION:
This study will assess the long-term protection offered by the new meningococcal vaccine GSK 134612 compared to Meningitec™ up to 4 years after vaccination of toddlers. Subjects were previously vaccinated at 12 to 23 months of age with GSK Biologicals' meningococcal vaccine GSK 134612 or Meningitec™. All subjects received at least one dose of Priorix-Tetra™. This extension phase starts 24 months after vaccination and the subjects who were vaccinated in the primary study will be enrolled in this extension study. No new subjects will be enrolled. The subjects will have a blood sample taken at 24, 36 and 48 months after primary vaccination.

At Year 4 subjects will be boosted with the same meningococcal vaccine as given in the primary study, i.e. either the new meningococcal vaccine GSK 134612 or Meningitec™. Blood samples will be taken 1 and 12 months after the booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the parent(s) or guardian(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* A male or female having completed the primary study 109670 and who was primed with the investigational or Meningitec™ vaccines.

Exclusion Criteria:

Exclusion criteria for persistence study entry (i.e. Month 24, 36 or 48):

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the subject's first visit.
* History of meningococcal disease.
* Administration of a meningococcal polysaccharide or a meningococcal polysaccharide conjugate vaccine outside of study 109670.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* Administration of immunoglobulins and/or blood products within the three months preceding the subjects first visit.
* Concurrently participating in another clinical study, within 30 days of study entry, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Bleeding disorders, such as thrombocytopenia, or subjects on anti-coagulant therapy.

Additional exclusion criteria for booster vaccination (to be checked at Month 48):

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to any vaccine containing diphtheria toxoid or non-toxic diphtheria toxin protein and/or tetanus toxoid.
* History of hypersensitivity after previous administration of Meningitec or the investigational vaccines in study 109670.
* Hypersensitivity to latex.
* Planned administration/ administration of a vaccine not foreseen by the protocol within one month before and 30 days after the booster dose.
* Previous vaccination with any component of the vaccines within the last month.
* History of any neurological disorder or seizures (one episode of febrile convulsion does not constitute an exclusion criteria).
* Major congenital defects or serious chronic illness.
* Acute disease at the time of vaccination.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2009-08-25 (Actual); Primary Completion 2009-12-16 (Actual); Study Completion 2012-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Finland (12):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Vesikari T, Forsten A, Bianco V, Van der Wielen M, Miller JM. Immunogenicity, Safety and Antibody Persistence of a Booster Dose of Quadrivalent Meningococcal ACWY-tetanus Toxoid Conjugate Vaccine Compared with Monovalent Meningococcal Serogroup C Vaccine Administered Four Years After Primary Vaccination Using the Same Vaccines. Pediatr Infect Dis J. 2015 Dec;34(12):e298-307. doi: 10.1097/INF.0000000000000897. PMID 26780033
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not all study participants returned in time for every study visit, but they were allowed to continue the study nonetheless. The number of participants who started each study period depends on the actual rate of return of the subjects.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Nimenrix Group: Subjects vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and who at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study.
- Meningitec Group: Subjects who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
Period: Year 2 Period
Arm/Group | Nimenrix Group | Meningitec Group
Started | 253 | 42
Completed | 253 | 42
Not Completed | 0 | 0
Period: Year 3 Period
Arm/Group | Nimenrix Group | Meningitec Group
Started | 273 | 47
Completed | 273 | 47
Not Completed | 0 | 0
Period: Year 4 Period
Arm/Group | Nimenrix Group | Meningitec Group
Started | 246 | 48
Completed | 246 | 48
Not Completed | 0 | 0
Period: Booster Period (Month 48- 49)
Arm/Group | Nimenrix Group | Meningitec Group
Started | 245 | 48
Completed | 244 | 47
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Year 5 Period
Arm/Group | Nimenrix Group | Meningitec Group
Started | 239 | 47
Completed | 239 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nimenrix Group (Y2 - Y 5): Subjects from Year 2, 3, 4, Month 49 and Year 5 period, vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and who at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study.
- Meningitec Group (Y 2- Y 5): Subjects from Year 2, 3, 4, Month 49 and Year 5 period, who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
- Total: Total of all reporting groups
Arm/Group | Nimenrix Group (Y2 - Y 5) | Meningitec Group (Y 2- Y 5) | Total
Number analyzed (Participants) | 1256 | 232 | 1488
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Note: The numbers analyzed in rows represent the number of subjects at the respective study periods.
  Months
    Year 2 Period: number analyzed (Participants) | 253 | 42 | 295
    Year 2 Period | 40.7 (1.87) | 41.1 (1.74) | 40.76 (1.85)
    Year 3 Period: number analyzed (Participants) | 273 | 47 | 320
    Year 3 Period | 49.0 (1.77) | 49.3 (2.09) | 49.04 (1.82)
    Year 4 Period: number analyzed (Participants) | 246 | 48 | 294
    Year 4 Period | 63.7 (1.81) | 63.9 (1.97) | 63.73 (1.84)
    Booster Period Month 49: number analyzed (Participants) | 245 | 48 | 293
    Booster Period Month 49 | 63.7 (1.81) | 63.9 (1.97) | 63.73 (1.84)
    Year 5 Period: number analyzed (Participants) | 239 | 47 | 286
    Year 5 Period | 72.9 (1.68) | 72.9 (1.83) | 72.9 (1.70)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Note: The numbers analyzed in rows represent the number of subjects at the respective study periods.
  Participants
    Year 2 Period: number analyzed (Participants) | 253 | 42 | 295
    Year 2 Period: Female | 120 | 20 | 140
    Year 2 Period: Male | 133 | 22 | 155
    Year 3 Period: number analyzed (Participants) | 273 | 47 | 320
    Year 3 Period: Female | 129 | 22 | 151
    Year 3 Period: Male | 144 | 25 | 169
    Year 4 Period: number analyzed (Participants) | 246 | 48 | 294
    Year 4 Period: Female | 120 | 22 | 142
    Year 4 Period: Male | 126 | 26 | 152
    Booster Period Month 49: number analyzed (Participants) | 245 | 48 | 293
    Booster Period Month 49: Female | 119 | 22 | 141
    Booster Period Month 49: Male | 126 | 26 | 152
    Year 5 Period: number analyzed (Participants) | 239 | 47 | 286
    Year 5 Period: Female | 116 | 22 | 138
    Year 5 Period: Male | 123 | 25 | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Note: The numbers analyzed in rows represent the number of subjects at the respective study periods.
  Participants
    Year 2 Period: number analyzed (Participants) | 253 | 42 | 295
    Year 2 Period: White - Caucasian / European heritage, n (%) | 252 | 42 | 294
    Year 2 Period: Other | 1 | 0 | 1
    Year 3 Period: number analyzed (Participants) | 273 | 47 | 320
    Year 3 Period: White - Caucasian / European heritage, n (%) | 271 | 47 | 318
    Year 3 Period: Other | 2 | 0 | 2
    Year 4 Period: number analyzed (Participants) | 246 | 48 | 294
    Year 4 Period: White - Caucasian / European heritage, n (%) | 245 | 47 | 292
    Year 4 Period: Other | 1 | 1 | 2
    Booster Period Month 49: number analyzed (Participants) | 245 | 48 | 293
    Booster Period Month 49: White - Caucasian / European heritage, n (%) | 244 | 47 | 291
    Booster Period Month 49: Other | 1 | 1 | 2
    Year 5 Period: number analyzed (Participants) | 239 | 47 | 286
    Year 5 Period: White - Caucasian / European heritage, n (%) | 238 | 46 | 284
    Year 5 Period: Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay /Activity (rSBA) Against Neisseria Meningitidis Serogroup A, C, W-135 and Y (Using Baby Rabbit Complement) Titres ≥ the Cut-off
Description: The cut-off value for the assay was greater than or equal to (≥) 1:8, as measured at the GlaxoSmithKline (GSK) laboratory.
Time Frame: At Month 24 post primary vaccination
Population: The analysis was performed on the According-To-Protocol cohort for persistence, which included all evaluable subjects who were eligible to participate in the primary study (109670) [NCT00474266], who complied with the protocol requirements and who had available assay results for at least one tested antigen.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group Y2: Subjects from Year 2 Period vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and who at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study.
- Meningitec Group Y2: Subjects from Year 2 Period who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 188 | 30
Participants
  rSBA-MenA [M24]: number analyzed (Participants) | 181 | 28
  rSBA-MenA [M24] | 177 | 23
  rSBA-MenC [M24]: number analyzed (Participants) | 186 | 29
  rSBA-MenC [M24] | 164 | 20
  rSBA-MenW-135 [M24]: number analyzed (Participants) | 188 | 29
  rSBA-MenW-135 [M24] | 186 | 17
  rSBA-MenY [M24] | 184 | 24

2. Primary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off value for the assay was ≥ 1:8. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group Y3: Subjects from Year 3 Period vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and who at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study.
- Meningitec Group Y3: Subjects from Year 3 Period who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 237 | 40
Participants
  rSBA-MenA [M36]: number analyzed (Participants) | 228 | 38
  rSBA-MenA [M36] | 224 | 32
  rSBA-MenC [M36]: number analyzed (Participants) | 235 | 39
  rSBA-MenC [M36] | 210 | 28
  rSBA-MenW-135 [M36]: number analyzed (Participants) | 236 | 39
  rSBA-MenW-135 [M36] | 232 | 22
  rSBA-MenY [M36] | 231 | 33

3. Primary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off value for the assay was ≥ 1:8. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 48 post primary vaccination
Population: The analysis was performed on the According-To-Protocol cohort for persistence, which included all evaluable subjects who were eligible to participate in the primary study (109670) [NCT00474266] , who complied with the protocol requirements and who had available assay results for at least one tested antigen.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group Y4: Subjects from Year 4 Period vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and who and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study.
- Meningitec Group Y4: Subjects from Year 4 Period who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 195 | 37
Participants
  rSBA-MenA [M48]: number analyzed (Participants) | 188 | 35
  rSBA-MenA [M48] | 185 | 29
  rSBA-MenC [M48]: number analyzed (Participants) | 194 | 36
  rSBA-MenC [M48] | 175 | 24
  rSBA-MenW-135 [M48]: number analyzed (Participants) | 194 | 36
  rSBA-MenW-135 [M48] | 192 | 22
  rSBA-MenY [M48] | 190 | 31

4. Primary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: The cut-off value for the assay was ≥ 1:8. The rSBA-MenA results for the Year 3 time point were obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 36 post-primary vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 262 | 46
Participants
  rSBA-MenA [M36] | 157 | 3
  rSBA-MenC [M36] | 94 | 6
  rSBA-MenW-135 [M36]: number analyzed (Participants) | 261 | 46
  rSBA-MenW-135 [M36] | 130 | 2
  rSBA-MenY [M36] | 141 | 6

5. Primary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: The cut-off value for the aasay was ≥ 1:8. The rSBA-MenA results for the Year 4 time point were obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 48 post-primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 225 | 45
Participants
  rSBA-MenA [M48]: number analyzed (Participants) | 224 | 45
  rSBA-MenA [M48] | 166 | 13
  rSBA-MenC [M48] | 91 | 16
  rSBA-MenW-135 [M48] | 111 | 7
  rSBA-MenY [M48] | 131 | 11

6. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBAMenY Titres ≥ the Cut-off
Description: The cut-off value for the assay was ≥ 1:128, as measured at the GlaxoSmithKline (GSK) laboratory.
Time Frame: At Month 24 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 188 | 30
Participants
  rSBA-MenA [M24]: number analyzed (Participants) | 181 | 28
  rSBA-MenA [M24] | 166 | 16
  rSBA-MenC [M24]: number analyzed (Participants) | 186 | 29
  rSBA-MenC [M24] | 90 | 14
  rSBA-MenW-135 [M24]: number analyzed (Participants) | 188 | 29
  rSBA-MenW-135 [M24] | 171 | 12
  rSBA-MenY [M24] | 154 | 20

7. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off value for the assay was ≥ 1:128. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 237 | 40
Participants
  rSBA-MenA [M36]: number analyzed (Participants) | 228 | 38
  rSBA-MenA [M36] | 207 | 23
  rSBA-MenC [M36]: number analyzed (Participants) | 235 | 39
  rSBA-MenC [M36] | 115 | 19
  rSBA-MenW-135 [M36]: number analyzed (Participants) | 236 | 39
  rSBA-MenW-135 [M36] | 211 | 16
  rSBA-MenY [M36] | 195 | 26

8. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off value for the assay was ≥ 1:128. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 48 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 195 | 37
Participants
  rSBA-MenA [M48]: number analyzed (Participants) | 188 | 35
  rSBA-MenA [M48] | 175 | 22
  rSBA-MenC [M48]: number analyzed (Participants) | 194 | 36
  rSBA-MenC [M48] | 97 | 18
  rSBA-MenW-135 [M48]: number analyzed (Participants) | 194 | 36
  rSBA-MenW-135 [M48] | 177 | 17
  rSBA-MenY [M48] | 163 | 25

9. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: The results for the assay were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres, as measured at the GlaxoSmithKline (GSK) laboratory
Time Frame: At Months 24 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 188 | 30
Titres
  rSBA-MenA [M24]: number analyzed (Participants) | 181 | 28
  rSBA-MenA [M24] | 420.3 [356.1 to 495.9] | 90.6 [46.2 to 177.9]
  rSBA-MenC [M24]: number analyzed (Participants) | 186 | 29
  rSBA-MenC [M24] | 98.1 [77.7 to 123.8] | 53.5 [25.5 to 112]
  rSBA-MenW-135 [M24]: number analyzed (Participants) | 188 | 29
  rSBA-MenW-135 [M24] | 396.9 [342 to 460.5] | 42.2 [18.5 to 96.4]
  rSBA-MenY [M24] | 396.6 [324 to 485.5] | 151.3 [69.2 to 330.6]

10. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: Results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 237 | 40
Titres
  rSBA-MenA [M36]: number analyzed (Participants) | 228 | 38
  rSBA-MenA [M36] | 415.3 [360.9 to 478] | 102.3 [59.6 to 175.4]
  rSBA-MenC [M36]: number analyzed (Participants) | 235 | 39
  rSBA-MenC [M36] | 104.2 [84.7 to 128.2] | 58.5 [31.7 to 107.9]
  rSBA-MenW-135 [M36]: number analyzed (Participants) | 236 | 39
  rSBA-MenW-135 [M36] | 372.4 [323.4 to 428.9] | 39.7 [19.5 to 80.5]
  rSBA-MenY [M36] | 405.4 [337.4 to 487.1] | 169.1 [89.6 to 319.1]

11. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: as for outcome 10
Time Frame: At Month 48 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 195 | 37
Titres
  rSBA-MenA [M48]: number analyzed (Participants) | 188 | 35
  rSBA-MenA [M48] | 437.1 [376.6 to 507.4] | 106.4 [58.8 to 192.4]
  rSBA-MenC [M48]: number analyzed (Participants) | 194 | 36
  rSBA-MenC [M48] | 105.4 [84.6 to 131.3] | 53.6 [27.1 to 105.8]
  rSBA-MenW-135 [M48]: number analyzed (Participants) | 194 | 36
  rSBA-MenW-135 [M48] | 398.2 [343.1 to 462.1] | 49.1 [23.5 to 102.5]
  rSBA-MenY [M48] | 411.1 [336.1 to 502.9] | 186.9 [98.1 to 355.8]

12. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBAMenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off for the assay was ≥ 1:128. rSBA-MenA, MenC, MenW and MenY results for the Year 3 time point obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 36 post-primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 262 | 46
Participants
  rSBA-MenA [M36] | 60 | 3
  rSBA-MenC [M36] | 23 | 3
  rSBA-MenW-135 [M36]: number analyzed (Participants) | 261 | 46
  rSBA-MenW-135 [M36] | 87 | 2
  rSBA-MenY [M36] | 75 | 2

13. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off value for the assay was ≥ 1:128. rSBA-MenA, MenC, MenW and MenY results for the Year 4 time point obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 48 post-primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 225 | 45
Participants
  rSBA-MenA [M48]: number analyzed (Participants) | 224 | 45
  rSBA-MenA [M48] | 134 | 12
  rSBA-MenC [M48] | 34 | 10
  rSBA-MenW-135 [M48] | 88 | 7
  rSBA-MenY [M48] | 91 | 9

14. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: Results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres. rSBA-MenA, MenC, MenW and MenY results for the Year 3 time point obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 36 post-primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 262 | 46
Titres
  rSBA-MenA [M36] | 19.3 [15.7 to 23.6] | 5.2 [3.8 to 6.9]
  rSBA-MenC [M36] | 9.8 [8.1 to 11.7] | 5.7 [4.2 to 7.7]
  rSBA-MenW-135 [M36]: number analyzed (Participants) | 261 | 46
  rSBA-MenW-135 [M36] | 24.9 [19.2 to 32.4] | 4.9 [3.7 to 6.7]
  rSBA-MenY [M36] | 22.3 [17.6 to 28.4] | 5.7 [4.2 to 7.8]

15. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: Results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres. rSBA-MenA, MenC, MenW and MenY results for the Year 4 time point were obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 48 post-primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 225 | 45
Titres
  rSBA-MenA [M48]: number analyzed (Participants) | 224 | 45
  rSBA-MenA [M48] | 107.3 [77.6 to 148.3] | 18.4 [8.5 to 39.7]
  rSBA-MenC [M48] | 12.3 [9.8 to 15.3] | 13.5 [7.4 to 24.5]
  rSBA-MenW-135 [M48] | 30.5 [22.4 to 41.5] | 8 [4.8 to 13.3]
  rSBA-MenY [M48] | 36.2 [27.1 to 48.4] | 10.4 [6 to 18]

16. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay/Activity Against Neisseria Meningitidis Serogroup A, C, W-135 and Y (Using Human Complement) Titres ≥ the Cut-off
Description: The cut-off values for the assay were ≥ 1:4 and 1:8, respectively. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 24 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 183 | 23
Participants
  hSBA-MenA [M24], ≥ 1:4 | 46 | 2
  hSBA-MenA [M24], ≥ 1:8 | 42 | 0
  hSBA-MenC [M24], ≥ 1:4: number analyzed (Participants) | 175 | 19
  hSBA-MenC [M24], ≥ 1:4 | 154 | 11
  hSBA-MenC [M24], ≥ 1:8: number analyzed (Participants) | 175 | 19
  hSBA-MenC [M24], ≥ 1:8 | 152 | 10
  hSBA-MenW-135 [M24], ≥ 1:4: number analyzed (Participants) | 180 | 23
  hSBA-MenW-135 [M24], ≥ 1:4 | 167 | 0
  hSBA-MenW-135 [M24], ≥ 1:8: number analyzed (Participants) | 180 | 23
  hSBA-MenW-135 [M24], ≥ 1:8 | 164 | 0
  hSBA-MenY [M24], ≥ 1:4: number analyzed (Participants) | 154 | 22
  hSBA-MenY [M24], ≥ 1:4 | 134 | 5
  hSBA-MenY [M24], ≥ 1:8: number analyzed (Participants) | 154 | 22
  hSBA-MenY [M24], ≥ 1:8 | 134 | 5

17. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay/Activity Against Neisseria Meningitidis Serogroup A, C, W-135 and Y (Using Human Complement) Titres ≥ the Cut-off
Description: The cut-off for the assay were ≥ 1:4 and 1:8. The analysis of this endpoint was performed by GSK.
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 258 | 35
Participants
  hSBA-MenA [M36], ≥ 1:4: number analyzed (Participants) | 251 | 31
  hSBA-MenA [M36], ≥ 1:4 | 95 | 5
  hSBA-MenA [M36], ≥ 1:8: number analyzed (Participants) | 251 | 31
  hSBA-MenA [M36], ≥ 1:8 | 90 | 4
  hSBA-MenC [M36], ≥ 1:4: number analyzed (Participants) | 253 | 31
  hSBA-MenC [M36], ≥ 1:4 | 204 | 13
  hSBA-MenC [M36], ≥ 1:8: number analyzed (Participants) | 253 | 31
  hSBA-MenC [M36], ≥ 1:8 | 198 | 13
  hSBA-MenW-135 [M36], ≥ 1:4: number analyzed (Participants) | 254 | 33
  hSBA-MenW-135 [M36], ≥ 1:4 | 209 | 2
  hSBA-MenW-135 [M36], ≥ 1:8: number analyzed (Participants) | 254 | 33
  hSBA-MenW-135 [M36], ≥ 1:8 | 209 | 2
  hSBA-MenY [M36], ≥ 1:4: number analyzed (Participants) | 250 | 33
  hSBA-MenY [M36], ≥ 1:4 | 184 | 6
  hSBA-MenY [M36], ≥ 1:8: number analyzed (Participants) | 250 | 33
  hSBA-MenY [M36], ≥ 1:8 | 180 | 6

18. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay/Activity Against Neisseria Meningitidis Serogroup A, C, W-135 and Y (Using Human Complement) Titres ≥ the Cut-off
Description: The cut-off for the assay were ≥ 1:4 and 1:8, as assessed by the GSK laboratory.
Time Frame: At Month 48 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 209 | 32
Participants
  hSBA-MenA [M48], ≥ 1:4: number analyzed (Participants) | 198 | 28
  hSBA-MenA [M48], ≥ 1:4 | 58 | 4
  hSBA-MenA [M48], ≥ 1:8: number analyzed (Participants) | 198 | 28
  hSBA-MenA [M48], ≥ 1:8 | 57 | 4
  hSBA-MenC [M48], ≥ 1:4 | 154 | 15
  hSBA-MenC [M48], ≥ 1:8 | 153 | 15
  hSBA-MenW-135 [M48], ≥ 1:4: number analyzed (Participants) | 165 | 26
  hSBA-MenW-135 [M48], ≥ 1:4 | 134 | 2
  hSBA-MenW-135 [M48], ≥ 1:8: number analyzed (Participants) | 165 | 26
  hSBA-MenW-135 [M48], ≥ 1:8 | 133 | 2
  hSBA-MenY [M48], ≥ 1:4: number analyzed (Participants) | 130 | 27
  hSBA-MenY [M48], ≥ 1:4 | 85 | 6
  hSBA-MenY [M48], ≥ 1:8: number analyzed (Participants) | 130 | 27
  hSBA-MenY [M48], ≥ 1:8 | 85 | 6

19. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres
Description: The results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres, as assessed by the GSK laboratory.
Time Frame: At Month 24 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 183 | 23
Titres
  hSBA-MenA [M24] | 3.8 [3.2 to 4.5] | 2.2 [1.9 to 2.4]
  hSBA-MenC [M24]: number analyzed (Participants) | 175 | 19
  hSBA-MenC [M24] | 50.2 [38.7 to 65.1] | 10.4 [4.7 to 22.8]
  hSBA-MenW-135 [M24]: number analyzed (Participants) | 180 | 23
  hSBA-MenW-135 [M24] | 77.7 [61.8 to 97.6] | 2 [2 to 2]
  hSBA-MenY [M24]: number analyzed (Participants) | 154 | 22
  hSBA-MenY [M24] | 58.1 [44.5 to 75.8] | 5 [2.2 to 11.1]

20. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres
Description: as for outcome 19
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 254 | 33
Titres
  hSBA-MenA [M36]: number analyzed (Participants) | 251 | 31
  hSBA-MenA [M36] | 5.8 [4.8 to 7] | 2.6 [2.1 to 3.3]
  hSBA-MenC [M36]: number analyzed (Participants) | 253 | 31
  hSBA-MenC [M36] | 37.8 [29.4 to 48.6] | 6.2 [3.7 to 10.3]
  hSBA-MenW-135 [M36] | 52 [41.4 to 65.2] | 2.4 [1.8 to 3.1]
  hSBA-MenY [M36]: number analyzed (Participants) | 250 | 33
  hSBA-MenY [M36] | 33.2 [25.9 to 42.5] | 4.1 [2.4 to 7.1]

21. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres
Description: The results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres, as measured by GSK.
Time Frame: At Month 48 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 209 | 32
Titres
  hSBA-MenA [M48]: number analyzed (Participants) | 198 | 28
  hSBA-MenA [M48] | 4.9 [4 to 6] | 2.9 [2 to 4]
  hSBA-MenC [M48] | 32 [23.8 to 43] | 11.3 [4.9 to 25.6]
  hSBA-MenW-135 [M48]: number analyzed (Participants) | 165 | 26
  hSBA-MenW-135 [M48] | 47.1 [35.7 to 62.2] | 2.6 [1.8 to 3.8]
  hSBA-MenY [M48]: number analyzed (Participants) | 130 | 27
  hSBA-MenY [M48] | 29.8 [20.2 to 44.1] | 4.4 [2.4 to 8.1]

22. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 0.3 microgram per milliliter (μg/mL) and ≥ 2.0 μg/mL, respectively, as measured at the GlaxoSmithKline (GSK) laboratory.
Time Frame: At Month 24 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 92 | 17
Participants
  Anti-PSA [M24], ≥ 0.3 | 50 | 5
  Anti-PSA [M24], ≥ 2.0 | 8 | 2
  Anti-PSC [M24], ≥ 0.3: number analyzed (Participants) | 89 | 16
  Anti-PSC [M24], ≥ 0.3 | 25 | 3
  Anti-PSC [M24], ≥ 2.0: number analyzed (Participants) | 89 | 16
  Anti-PSC [M24], ≥ 2.0 | 0 | 0
  Anti-PSW-135 [M24], ≥ 0.3: number analyzed (Participants) | 86 | 16
  Anti-PSW-135 [M24], ≥ 0.3 | 56 | 0
  Anti-PSW-135 [M24], ≥ 2.0: number analyzed (Participants) | 86 | 16
  Anti-PSW-135 [M24], ≥ 2.0 | 8 | 0
  Anti-PSY [M24], ≥ 0.3: number analyzed (Participants) | 89 | 17
  Anti-PSY [M24], ≥ 0.3 | 72 | 0
  Anti-PSY [M24], ≥ 2.0: number analyzed (Participants) | 89 | 17
  Anti-PSY [M24], ≥ 2.0 | 25 | 0

23. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 0.3 μg/mL and ≥ 2.0 μg/mL, respectively, as measured by the GSK laboratory.
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 114 | 21
Participants
  Anti-PSA [M36], ≥ 0.3 | 61 | 6
  Anti-PSA [M36], ≥ 2.0 | 10 | 2
  Anti-PSC [M36], ≥ 0.3: number analyzed (Participants) | 111 | 20
  Anti-PSC [M36], ≥ 0.3 | 28 | 4
  Anti-PSC [M36], ≥ 2.0: number analyzed (Participants) | 111 | 20
  Anti-PSC [M36], ≥ 2.0 | 0 | 0
  Anti-PSW-135 [M36], ≥ 0.3: number analyzed (Participants) | 106 | 20
  Anti-PSW-135 [M36], ≥ 0.3 | 68 | 0
  Anti-PSW-135 [M36], ≥ 2.0: number analyzed (Participants) | 106 | 20
  Anti-PSW-135 [M36], ≥ 2.0 | 11 | 0
  Anti-PSY [M36], ≥ 0.3: number analyzed (Participants) | 110 | 21
  Anti-PSY [M36], ≥ 0.3 | 89 | 1
  Anti-PSY [M36], ≥ 2.0: number analyzed (Participants) | 110 | 21
  Anti-PSY [M36], ≥ 2.0 | 33 | 0

24. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 0.3 μg/mL and ≥ 2.0 μg/mL, respectively, as measured by GSK.
Time Frame: At Month 48 post primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 93 | 20
Participants
  Anti-PSA [M48], ≥ 0.3 | 50 | 5
  Anti-PSA [M48], ≥ 2.0 | 9 | 2
  Anti-PSC [M48], ≥ 0.3: number analyzed (Participants) | 91 | 19
  Anti-PSC [M48], ≥ 0.3 | 21 | 3
  Anti-PSC [M48], ≥ 2.0: number analyzed (Participants) | 91 | 19
  Anti-PSC [M48], ≥ 2.0 | 0 | 0
  Anti-PSW-135 [M48], ≥ 0.3: number analyzed (Participants) | 86 | 19
  Anti-PSW-135 [M48], ≥ 0.3 | 55 | 0
  Anti-PSW-135 [M48], ≥ 2.0: number analyzed (Participants) | 86 | 19
  Anti-PSW-135 [M48], ≥ 2.0 | 8 | 0
  Anti-PSY [M48], ≥ 0.3: number analyzed (Participants) | 90 | 20
  Anti-PSY [M48], ≥ 0.3 | 73 | 1
  Anti-PSY [M48], ≥ 2.0: number analyzed (Participants) | 90 | 20
  Anti-PSY [M48], ≥ 2.0 | 26 | 0

25. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: The results were tabulated as geometric mean antibody concentration calculated on all subjects, expressed in μg/mL, as measured at the GlaxoSmithKline (GSK) laboratory.
Time Frame: At Month 24 post primary dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 92 | 17
μg/mL
  Anti-PSA [M24] | 0.4 [0.32 to 0.5] | 0.28 [0.16 to 0.49]
  Anti-PSC [M24]: number analyzed (Participants) | 89 | 16
  Anti-PSC [M24] | 0.22 [0.19 to 0.25] | 0.19 [0.14 to 0.27]
  Anti-PSW-135 [M24]: number analyzed (Participants) | 86 | 16
  Anti-PSW-135 [M24] | 0.47 [0.37 to 0.59] | 0.15 [0.15 to 0.15]
  Anti-PSY [M24]: number analyzed (Participants) | 89 | 17
  Anti-PSY [M24] | 0.85 [0.65 to 1.12] | 0.15 [0.15 to 0.15]

26. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: The results were tabulated as geometric mean antibody concentration calculated on all subjects, expresssed in μg/mL, as measured by GSK.
Time Frame: At Month 36 post primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 114 | 21
μg/mL
  Anti-PSA [M36] | 0.39 [0.32 to 0.48] | 0.27 [0.17 to 0.43]
  Anti-PSC [M36]: number analyzed (Participants) | 111 | 20
  Anti-PSC [M36] | 0.21 [0.19 to 0.24] | 0.19 [0.15 to 0.25]
  Anti-PSW-135 [M36]: number analyzed (Participants) | 106 | 20
  Anti-PSW-135 [M36] | 0.48 [0.39 to 0.59] | 0.15 [0.15 to 0.15]
  Anti-PSY [M36]: number analyzed (Participants) | 110 | 21
  Anti-PSY [M36] | 0.89 [0.7 to 1.14] | 0.16 [0.14 to 0.17]

27. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: as for outcome 26
Time Frame: At Month 48 post primary dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 93 | 20
μg/mL
  Anti-PSA [M48] | 0.39 [0.31 to 0.5] | 0.26 [0.16 to 0.42]
  Anti-PSC [M48]: number analyzed (Participants) | 91 | 19
  Anti-PSC [M48] | 0.2 [0.18 to 0.23] | 0.19 [0.14 to 0.25]
  Anti-PSW-135 [M48]: number analyzed (Participants) | 86 | 19
  Anti-PSW-135 [M48] | 0.46 [0.37 to 0.58] | 0.15 [0.15 to 0.15]
  Anti-PSY [M48]: number analyzed (Participants) | 90 | 20
  Anti-PSY [M48] | 0.89 [0.68 to 1.15] | 0.16 [0.14 to 0.17]

28. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 0.3 μg/mL and ≥ 0.2 μg/mL. Anti-PS results for the Year 3 time point were obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 36 post-primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 130 | 26
Participants
  Anti-PSA [M36], ≥ 0.3 | 128 | 20
  Anti-PSA [M36], ≥ 2.0 | 27 | 3
  Anti-PSC [M36], ≥ 0.3: number analyzed (Participants) | 119 | 25
  Anti-PSC [M36], ≥ 0.3 | 37 | 5
  Anti-PSC [M36], ≥ 2.0: number analyzed (Participants) | 119 | 25
  Anti-PSC [M36], ≥ 2.0 | 2 | 1
  Anti-PSW-135 [M36], ≥ 0.3: number analyzed (Participants) | 122 | 25
  Anti-PSW-135 [M36], ≥ 0.3 | 117 | 11
  Anti-PSW-135 [M36], ≥ 2.0: number analyzed (Participants) | 122 | 25
  Anti-PSW-135 [M36], ≥ 2.0 | 13 | 0
  Anti-PSY [M36], ≥ 0.3: number analyzed (Participants) | 104 | 22
  Anti-PSY [M36], ≥ 0.3 | 102 | 19
  Anti-PSY [M36], ≥ 2.0: number analyzed (Participants) | 104 | 22
  Anti-PSY [M36], ≥ 2.0 | 19 | 1

29. Secondary Outcome: Number of Subjects With Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off Values
Description: The cut-off values for the assay were ≥ 0.3 μg/mL and ≥ 2.0 μg/mL, respectively. Anti-PS results for the Year 4 time point were obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 48 post-primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 56 | 22
Participants
  Anti-PSA [M48], ≥ 0.3: number analyzed (Participants) | 53 | 22
  Anti-PSA [M48], ≥ 0.3 | 53 | 20
  Anti-PSA [M48], ≥ 2.0: number analyzed (Participants) | 53 | 22
  Anti-PSA [M48], ≥ 2.0 | 26 | 9
  Anti-PSC [M48], ≥ 0.3: number analyzed (Participants) | 56 | 21
  Anti-PSC [M48], ≥ 0.3 | 16 | 7
  Anti-PSC [M48], ≥ 2.0: number analyzed (Participants) | 56 | 21
  Anti-PSC [M48], ≥ 2.0 | 3 | 3
  Anti-PSW-135 [M48], ≥ 0.3 | 56 | 17
  Anti-PSW-135 [M48], ≥ 2.0 | 5 | 0
  Anti-PSY [M48], ≥ 0.3: number analyzed (Participants) | 50 | 20
  Anti-PSY [M48], ≥ 0.3 | 48 | 18
  Anti-PSY [M48], ≥ 2.0: number analyzed (Participants) | 50 | 20
  Anti-PSY [M48], ≥ 2.0 | 7 | 3

30. Secondary Outcome: Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: The results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in μg/mL. Anti-PS results for the Year 3 time point were obtained by re-testing the samples in parallel at Public Health England (PHE). Results were tabulated as geometric mean antibody concentration calculated on all subjects, expressed in μg/mL.
Time Frame: At Month 36 post-primary vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 130 | 26
μg/mL
  Anti-PSA [M36] | 1.16 [1.01 to 1.34] | 0.69 [0.45 to 1.06]
  Anti-PSC [M36]: number analyzed (Participants) | 119 | 25
  Anti-PSC [M36] | 0.22 [0.2 to 0.25] | 0.19 [0.15 to 0.25]
  Anti-PSW-135 [M36]: number analyzed (Participants) | 122 | 25
  Anti-PSW-135 [M36] | 0.78 [0.69 to 0.89] | 0.24 [0.19 to 0.3]
  Anti-PSY [M36]: number analyzed (Participants) | 104 | 22
  Anti-PSY [M36] | 1.12 [0.97 to 1.29] | 0.52 [0.37 to 0.72]

31. Secondary Outcome: Anti-polysaccharide A (Anti-PSA), Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: The results were tabulated as geometric mean antibody concentration calculated on all subjects, expressed in μg/mL. Anti-PS results for the Year 4 time point obtained by re-testing the samples in parallel at Public Health England (PHE).
Time Frame: At Month 48 post-primary vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 56 | 22
μg/mL
  Anti-PSA [M48]: number analyzed (Participants) | 53 | 22
  Anti-PSA [M48] | 2.05 [1.61 to 2.61] | 1.65 [0.97 to 2.83]
  Anti-PSC [M48]: number analyzed (Participants) | 56 | 21
  Anti-PSC [M48] | 0.25 [0.19 to 0.33] | 0.31 [0.18 to 0.54]
  Anti-PSW-135 [M48] | 0.85 [0.73 to 0.98] | 0.35 [0.28 to 0.46]
  Anti-PSY [M48]: number analyzed (Participants) | 50 | 20
  Anti-PSY [M48] | 0.77 [0.63 to 0.93] | 0.83 [0.54 to 1.28]

32. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres ≥ the Cut-off
Description: The cut-off values for the assay were 1:8 and 1:128, as measured by the PHE laboratory.
Time Frame: At one month (Month 49) post booster dose
Population: The analysis was performed on the Booster According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the booster vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group Month 49: Subjects from Booster Group vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group).
- Meningitec Booster Group (Month 49): Subjects from Booster Group who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 215 | 43
Participants
  rSBA-MenA [M49], ≥ 1:8: number analyzed (Participants) | 214 | 43
  rSBA-MenA [M49], ≥ 1:8 | 214 | 9
  rSBA-MenA [M49], ≥ 1:128: number analyzed (Participants) | 214 | 43
  rSBA-MenA [M49], ≥ 1:128 | 214 | 8
  rSBA-MenC [M49], ≥ 1:8 | 215 | 43
  rSBA-MenC [M49], ≥ 1:128 | 215 | 43
  rSBA-MenW-135 [M49], ≥ 1:8 | 215 | 8
  rSBA-MenW-135 [M49], ≥ 1:128 | 215 | 7
  rSBA-MenY [M49], ≥ 1:8 | 215 | 14
  rSBA-MenY [M49], ≥ 1:128 | 215 | 14

33. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres Above the Cut-off Values
Description: The cut off values for the assay were 1:8 and 1:128, as measured by the PHE laboratory.
Time Frame: At 12 months (Month 60) post booster dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Nimenrix Group Y5: Subjects from Year 5 Period vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and who at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study
- Meningitec Group Y5: Subjects from Year 5 Period who received Meningitec vaccine in the primary vaccination study 109670 [NCT00474266] (Priorix-Tetra Group and Meningitec Group) and at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study, as the only treatment administered after the primary study.
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 231 | 46
Participants
  rSBA-MenA [M60], ≥ 1:8 | 231 | 3
  rSBA-MenA [M60], ≥ 1:128 | 229 | 3
  rSBA-MenC [M60], ≥ 1:8 | 225 | 45
  rSBA-MenC [M60], ≥ 1:128 | 181 | 40
  rSBA-MenW-135 [M60], ≥ 1:8 | 231 | 2
  rSBA-MenW-135 [M60], ≥ 1:128 | 229 | 2
  rSBA-MenY [M60], ≥ 1:8 | 231 | 11
  rSBA-MenY [M60], ≥ 1:128 | 229 | 11

34. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: Results were tabulated as geometric mean antibody titre calculated on all subjects, expressed in titres, as measured by the PHE laboratory.
Time Frame: At one month (Month 49) post booster dose
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 215 | 43
Titres
  rSBA-MenA [M49]: number analyzed (Participants) | 214 | 43
  rSBA-MenA [M49] | 7173.3 [6389.2 to 8053.5] | 10.7 [5.6 to 20.4]
  rSBA-MenC [M49] | 4511.9 [3935.9 to 5172.3] | 3718.4 [2596 to 5326]
  rSBA-MenW-135 [M49] | 10949.7 [9531.4 to 12579.1] | 9.6 [5.3 to 17.3]
  rSBA-MenY [M49] | 4585.3 [4128.6 to 5092.5] | 15 [8 to 28]

35. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titres
Description: Results were tabulated as geometric mean antibody titre (GMT) calculated on all subjects, as measured by the PHE laboratory.
Time Frame: At 12 months (Month 60) post booster dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 231 | 46
Titres
  rSBA-MenA [M60] | 978.9 [860.2 to 1114] | 5.4 [3.8 to 7.6]
  rSBA-MenC [M60] | 226.4 [183.7 to 279] | 320.9 [201.1 to 512.2]
  rSBA-MenW-135 [M60] | 1390.7 [1203.2 to 1607.3] | 4.7 [3.8 to 5.7]
  rSBA-MenY [M60] | 1071.1 [924.9 to 1240.5] | 13.4 [6.9 to 25.8]

36. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres Above the Cut-off Values
Description: The cut off values for the assay were ≥ 1:4 and ≥ 1:8 respectively, as measured by GSK.
Time Frame: At one month (Month 49) post booster dose
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 209 | 33
Participants
  hSBA-MenA [M49], ≥ 1:4: number analyzed (Participants) | 202 | 28
  hSBA-MenA [M49], ≥ 1:4 | 201 | 4
  hSBA-MenA [M49], ≥ 1:8: number analyzed (Participants) | 202 | 28
  hSBA-MenA [M49], ≥ 1:8 | 201 | 4
  hSBA-MenC [M49], ≥ 1:4 | 209 | 33
  hSBA-MenC [M49], ≥ 1:8 | 209 | 33
  hSBA-MenW-135 [M49], ≥ 1:4: number analyzed (Participants) | 192 | 25
  hSBA-MenW-135 [M49], ≥ 1:4 | 192 | 1
  hSBA-MenW-135 [M49], ≥ 1:8: number analyzed (Participants) | 192 | 25
  hSBA-MenW-135 [M49], ≥ 1:8 | 192 | 1
  hSBA-MenY [M49], ≥ 1:4: number analyzed (Participants) | 173 | 25
  hSBA-MenY [M49], ≥ 1:4 | 173 | 6
  hSBA-MenY [M49], ≥ 1:8: number analyzed (Participants) | 173 | 25
  hSBA-MenY [M49], ≥ 1:8 | 173 | 6

37. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres Above the Cut-off Values
Description: The cut off values for the assay were ≥ 1:4 and ≥ 1:8, respectively, as measured by GSK.
Time Frame: At 12 months (Month 60) post booster dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 228 | 33
Participants
  hSBA-MenA [M60], ≥ 1:4: number analyzed (Participants) | 221 | 28
  hSBA-MenA [M60], ≥ 1:4 | 211 | 3
  hSBA-MenA [M60], ≥ 1:8: number analyzed (Participants) | 221 | 28
  hSBA-MenA [M60], ≥ 1:8 | 211 | 3
  hSBA-MenC [M60], ≥ 1:4 | 228 | 33
  hSBA-MenC [M60], ≥ 1:8 | 228 | 33
  hSBA-MenW-135 [M60], ≥ 1:4: number analyzed (Participants) | 218 | 31
  hSBA-MenW-135 [M60], ≥ 1:4 | 218 | 5
  hSBA-MenW-135 [M60], ≥ 1:8: number analyzed (Participants) | 218 | 31
  hSBA-MenW-135 [M60], ≥ 1:8 | 218 | 5
  hSBA-MenY [M60], ≥ 1:4: number analyzed (Participants) | 206 | 31
  hSBA-MenY [M60], ≥ 1:4 | 206 | 10
  hSBA-MenY [M60], ≥ 1:8: number analyzed (Participants) | 206 | 31
  hSBA-MenY [M60], ≥ 1:8 | 206 | 10

38. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres
Description: The results were tabulated as geometric mean antibody titre (GMT) calculated on all subjects, expressed in titres, as measured by GSK.
Time Frame: At one month (Month 49) post booster dose
Population: The analysis was performed on the Booster According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month after the booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 209 | 33
Titres
  hSBA-MenA [M49]: number analyzed (Participants) | 202 | 28
  hSBA-MenA [M49] | 1343.2 [1119.3 to 1612] | 2.8 [2 to 3.8]
  hSBA-MenC [M49] | 15831.4 [13625.8 to 18394] | 8646.1 [5886.6 to 12699.3]
  hSBA-MenW-135 [M49]: number analyzed (Participants) | 192 | 25
  hSBA-MenW-135 [M49] | 14411.2 [12971.8 to 16010.2] | 2.3 [1.7 to 3.3]
  hSBA-MenY [M49]: number analyzed (Participants) | 173 | 25
  hSBA-MenY [M49] | 6775.5 [5961.3 to 7700.9] | 4.9 [2.4 to 9.8]

39. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Titres
Description: as for outcome 38
Time Frame: At 12 months (Month 60) post booster dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 228 | 33
Titres
  hSBA-MenA [M60]: number analyzed (Participants) | 221 | 28
  hSBA-MenA [M60] | 88 [73.6 to 105.1] | 2.5 [1.9 to 3.2]
  hSBA-MenC [M60] | 1342.3 [1134.6 to 1588.1] | 931.1 [572.8 to 1513.4]
  hSBA-MenW-135 [M60]: number analyzed (Participants) | 218 | 31
  hSBA-MenW-135 [M60] | 2196.6 [1955.7 to 2467.2] | 3.4 [2.2 to 5.4]
  hSBA-MenY [M60]: number analyzed (Participants) | 206 | 31
  hSBA-MenY [M60] | 1110.8 [987.5 to 1249.6] | 7.5 [3.6 to 15.7]

40. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY Above the Cut-off Values
Description: The cut-off values for the assay were 0.3 μg/mL and 2.0 μg/mL, as measured by the PHE laboratory.
Time Frame: At one month (Month 49) post booster dose
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 70 | 19
Participants
  Anti-PSA [M49], ≥ 0.3: number analyzed (Participants) | 67 | 15
  Anti-PSA [M49], ≥ 0.3 | 67 | 15
  Anti-PSA [M49], ≥ 2.0: number analyzed (Participants) | 67 | 15
  Anti-PSA [M49], ≥ 2.0 | 66 | 6
  Anti-PSC [M49], ≥ 0.3: number analyzed (Participants) | 70 | 18
  Anti-PSC [M49], ≥ 0.3 | 70 | 18
  Anti-PSC [M49], ≥ 2.0: number analyzed (Participants) | 70 | 18
  Anti-PSC [M49], ≥ 2.0 | 67 | 18
  Anti-PSW-135 [M49], ≥ 0.3: number analyzed (Participants) | 69 | 19
  Anti-PSW-135 [M49], ≥ 0.3 | 69 | 13
  Anti-PSW-135 [M49], ≥ 2.0: number analyzed (Participants) | 69 | 19
  Anti-PSW-135 [M49], ≥ 2.0 | 69 | 0
  Anti-PSY [M49], ≥ 0.3: number analyzed (Participants) | 64 | 10
  Anti-PSY [M49], ≥ 0.3 | 63 | 9
  Anti-PSY [M49], ≥ 2.0: number analyzed (Participants) | 64 | 10
  Anti-PSY [M49], ≥ 2.0 | 63 | 0

41. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY ≥ the Cut-off Values
Description: The cut-off for the assay were 0.3 μg/mL and 2.0 μg/mL, as measured by the PHE laboratory.
Time Frame: At 12 months (Month 60) post booster dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 98 | 22
Participants
  Anti-PSA [M60], ≥ 0.3 | 98 | 22
  Anti-PSA [M60], ≥ 2.0 | 82 | 5
  Anti-PSC [M60], ≥ 0.3: number analyzed (Participants) | 85 | 14
  Anti-PSC [M60], ≥ 0.3 | 85 | 13
  Anti-PSC [M60], ≥ 2.0: number analyzed (Participants) | 85 | 14
  Anti-PSC [M60], ≥ 2.0 | 38 | 10
  Anti-PSW-135 [M60], ≥ 0.3 | 98 | 8
  Anti-PSW-135 [M60], ≥ 2.0 | 98 | 0
  Anti-PSY [M60], ≥ 0.3: number analyzed (Participants) | 86 | 12
  Anti-PSY [M60], ≥ 0.3 | 85 | 12
  Anti-PSY [M60], ≥ 2.0: number analyzed (Participants) | 86 | 12
  Anti-PSY [M60], ≥ 2.0 | 85 | 6

42. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: The results were tabulated as geometric mean antibody concentration calculated on all subjects, expressed in μg/mL, as measured by the PHE laboratory.
Time Frame: At one month (Month 49) post booster dose
Population: as for outcome 32
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 70 | 19
μg/mL
  Anti-PSA [M49]: number analyzed (Participants) | 67 | 15
  Anti-PSA [M49] | 12.61 [10.39 to 15.29] | 1.76 [1.1 to 2.81]
  Anti-PSC [M49]: number analyzed (Participants) | 70 | 18
  Anti-PSC [M49] | 8.64 [7.18 to 10.4] | 13.07 [9.09 to 18.8]
  Anti-PSW-135 [M49]: number analyzed (Participants) | 69 | 19
  Anti-PSW-135 [M49] | 59.06 [49.26 to 70.81] | 0.34 [0.24 to 0.48]
  Anti-PSY [M49]: number analyzed (Participants) | 64 | 10
  Anti-PSY [M49] | 38.85 [30.2 to 49.98] | 0.56 [0.35 to 0.89]

43. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW, and Anti-PSY Antibody Concentrations
Description: as for outcome 42
Time Frame: At 12 months (Month 60) post booster dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 98 | 22
μg/mL
  Anti-PSA [M60] | 4.22 [3.64 to 4.88] | 1.41 [1.09 to 1.82]
  Anti-PSC [M60]: number analyzed (Participants) | 85 | 14
  Anti-PSC [M60] | 1.81 [1.56 to 2.11] | 2.93 [1.47 to 5.86]
  Anti-PSW-135 [M60] | 9.44 [8.29 to 10.74] | 0.26 [0.18 to 0.37]
  Anti-PSY [M60]: number analyzed (Participants) | 86 | 12
  Anti-PSY [M60] | 10.31 [8.64 to 12.29] | 2.24 [1.25 to 4.02]

44. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 8-day period (Days 0-7) after booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary study (109670) [NCT00474266], with a booster vaccine administration documented and with their symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 244 | 47
Participants
  Any pain | 149 | 23
  Any Redness | 90 | 17
  Any Swelling | 70 | 11

45. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, irritability, loss of appetite, temperature (measured orally). Any was defined as occurrence of any general symptoms, regardless of their intensity grade or their relationship to vaccination
Time Frame: During the 8-day period (Days 0-7) after the booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary study (109670) [NCT00474266], with a booster vaccine administration documented, and with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 244 | 47
Participants
  Any drowsiness | 41 | 10
  Any irritability: number analyzed (Participants) | 243 | 47
  Any irritability | 40 | 11
  Any loss of appetite: number analyzed (Participants) | 243 | 47
  Any loss of appetite | 31 | 8
  Any temperature (orally, ≥ 37.5°C): number analyzed (Participants) | 243 | 47
  Any temperature (orally, ≥ 37.5°C) | 16 | 1

46. Secondary Outcome: Number of Subjects Reporting Any Adverse Events (AEs)
Description: Any was defined as the occurrence of any adverse event regardless of intensity grade or relation to vaccination. An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regard-less of intensity grade or relation to vaccination.
Time Frame: During the 31-day period (Days 0-30) after booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary study (109670) [NCT00474266], with a booster vaccine administration documented, and with their symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 245 | 48
Participants | 106 | 18

47. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity.
Time Frame: At Month 24 post primary dose
Population: The analysis was performed on the Total cohort for each persistence time point, which included all vaccinated subjects in the primary study (109670) [NCT00474266], who came back to the visit at the considered time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y2 | Meningitec Group Y2
Number analyzed (Participants) | 253 | 42
Participants | 0 | 0

48. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: as for outcome 47
Time Frame: At Month 36
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y3 | Meningitec Group Y3
Number analyzed (Participants) | 273 | 47
Participants | 0 | 0

49. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: as for outcome 47
Time Frame: At Month 48
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y4 | Meningitec Group Y4
Number analyzed (Participants) | 246 | 48
Participants | 0 | 0

50. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: as for outcome 47
Time Frame: From month 48 to month 49 (post booster follow up period)
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects in the primary study (109670) [NCT00474266], with a booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Month 49 | Meningitec Booster Group (Month 49)
Number analyzed (Participants) | 245 | 48
Participants | 2 | 0

51. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: as for outcome 47
Time Frame: From month 49 to month 60
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix Group Y5 | Meningitec Group Y5
Number analyzed (Participants) | 239 | 47
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 8-day period (Days 0-7) after booster vaccination. Unsolicited symptoms: during the 31-day period (Days 0-30) after booster vaccination. SAEs: during the 31-day period (Days 0-30) following booster vaccination.
Description: The solicited local and general symptoms were only collected for those subjects who filled-in their symptom sheets.
Groups:
- Nimenrix Group: Subjects vaccinated with Nimenrix vaccine in the primary study 109670 [NCT00474266] (Nimenrix+ Priorix-Tetra Group and Nimenrix Group) and and who at Year 4 received a booster dose with the same meningococcal vaccine as given in the primary study.
Arm/Group | Nimenrix Group | Meningitec Group
All-Cause Mortality (participants affected / at risk) | 0/245 | 0/48
Serious Adverse Events (participants affected / at risk) | 2/245 | 0/48
Other Adverse Events (participants affected / at risk) | 190/245 | 39/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix Group (N=245) | Meningitec Group (N=48)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix Group (N=245) | Meningitec Group (N=48)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 31 (31) | 8 (8)
Erythema (Skin and subcutaneous tissue disorders) | 90 (90) | 17 (17)
Headache (Nervous system disorders) | 5 (6) | 3 (4)
Irritability (Psychiatric disorders) | 40 (40) | 11 (11)
Nasopharyngitis (Infections and infestations) | 13 (14) | 1 (1)
Pain (General disorders) | 149 (149) | 23 (23)
Pyrexia (General disorders) | 23 (23) | 4 (4)
Somnolence (Nervous system disorders) | 41 (41) | 10 (10)
Swelling (General disorders) | 70 (70) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.